CLINICAL TRIAL: NCT05299658
Title: An Open-Label Extension for the Phase 2, Randomised, Double-Blind, Placebo-Controlled Study in Early Symptomatic Amyotrophic Lateral Sclerosis Patients on Stable Background Therapy to Assess Bioenergetic Catalysis With CNM-Au8 to Slow Disease Progression in ALS
Brief Title: An Open-Label Extension for the Phase 2 Study in Early Symptomatic Amyotrophic Lateral Sclerosis Patients on Stable Background Therapy to Assess Bioenergetic Catalysis With CNM-Au8 to Slow Disease Progression in ALS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clene Nanomedicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNMAu8.205 OLE
Expanded Access: NCT04081714 (Temporarily not available)
Record Dates: First submitted 2022-03-08; First posted 2022-03-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Open-label extension
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Open-label extension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label extension (Experimental): This is an unblinded open-label extension, all participants will be on active drug.
  Interventions: Drug: CNMAu8

INTERVENTIONS:
Drug: CNMAu8 — CNM-Au8 is an aqueous suspension of clean surfaced faceted nanocrystals consisting of gold atoms self-organized into crystals of various geometrical shapes (hexagonal bi-pyramid, pentagonal bi-pyramid, tetrahedron, decahedron, planar spheroids). Those choosing to participate in the OLE period will orally receive 30 mg of CNM-Au8, once daily.

SUMMARY:
This is an optional open-label extension to participants that have completed the clinical trial CNMAu8.205.

DETAILED DESCRIPTION:
A forty-eight (48) week optional open-label extension period (Open- Label Period), which may be extended by 12-week increments until discontinued by the Sponsor for participants that have completed protocol CNMAu8.205.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have completed the randomized placebo-controlled Treatment Period without compliance issues.
2. Able to understand and give written informed consent to participate in the open-label extension.
3. If referred from a third party (neurologist or a State based ALS organisation), participant agrees to maintain transfer of care to a neurologist participating in the study.

Exclusion Criteria:

1. Lack of treatment compliance during the randomized placebo controlled Treatment Period.
2. Positive pregnancy test at the Week 36 visit, or, females who plan to get pregnant during the course of this extension or within 6 months of the end of this extension.
3. Based on the investigator's judgment, patients who may have difficulty complying with the protocol and/or any study procedures.
4. Patient with clinically significant abnormalities in haematology, blood chemistry, ECG, or physical examination identified during the W36 visit which according to Investigator may interfere with continued participation.
5. Patients with clinically significant hepatic or renal dysfunction or clinical laboratory findings that would limit the interpretability of change in liver or kidney function, or those with low platelet counts (< 150 x 10^9 per liter) or eosinophilia (absolute eosinophil count of ≥ 500 eosinophils per microliter) at the Week 36 visit.
6. Patient is considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Safety measures | Up to an estimated 96 weeks.
  Safety endpoints include incidence of treatment-emergent AEs, drug-related AEs, deaths, SAEs, and AEs leading to discontinuation from the study. Changes from baseline (Week 36 of the placebo controlled phase) in clinical laboratory results, physical examination findings, vital signs, ECGs, and C-SSRS will be summarized descriptively by group and timepoint.
Electromyography measures | Up to an estimated 96 weeks.
  Mean change in the average difference between active treatment and placebo from Baseline through End of Study for the MUNIXscore(4), which is the sum of the respective MUNIX values for the Abductor Digiti Minimi (ADM), Abductor Pollicis Brevis (APB), Biceps Brachii (BB), and Tibialis Anterior (TA).

OTHER OUTCOMES:
MScanFit MUNE | Up to an estimated 96 weeks.
  Mean change in the average difference between active treatment and placebo from Baseline through Week 36 (overall difference at all time points) as measured by MScanFit MUNE (Jacobsen et al., 2017) of the APB in the least clinically affected hand. The baseline average will be indexed to 100%, and changes at Week 12, 24 and Week 36 will be calculated as the percent change from the Baseline index of 100%.
MUSIX | Up to an estimated 96 weeks.
  Mean change in the average difference between active treatment and placebo from Baseline through Week 36 for the MUSIXscore(4) (Neuwirth et al., 2015), which is the mean of the respective MUSIX values for the ADM, APB, BB, and TA. The average baseline mean values will be indexed to 100%. Changes will be calculated as the percent change from the Baseline index of 100%. baseline average will be indexed to 100%, and changes at Week 12, 24 and Week 36 will be calculated as the percent change from the Baseline index of 100%.
Spilt Hand Index | Up to an estimated 96 weeks.
  Mean change in the average difference between active treatment and placebo from Baseline through Week 36 for the Split Hand Index (SI) (Menon et al., 2013), defined as the first dorsal interosseous (FDI)Peak CMAP Amplitude * APBPeak CMAP Amplitude/ADMPeak CMAP Amplitude.
Neurophysiological index | Up to an estimated 96 weeks.
  Mean change in the average difference between active treatment and placebo from Baseline through Week 36 for the Neurophysiological Index (NPI) of the ADM (Cheah et al., 2011), defined as the ulnar nerve (ADMCMAP Peak Amplitude / ADMDistal Motor Latency) * ADMF-Wave (%).

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Concord Hospital, Concord, New South Wales
  - Neuroscience Research Australia, Randwick, New South Wales

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vucic S, Menon P, Huynh W, Mahoney C, Ho KS, Hartford A, Rynders A, Evan J, Evan J, Ligozio S, Glanzman R, Hotchkin MT, Kiernan MC. Efficacy and safety of CNM-Au8 in amyotrophic lateral sclerosis (RESCUE-ALS study): a phase 2, randomised, double-blind, placebo-controlled trial and open label extension. EClinicalMedicine. 2023 Jun 8;60:102036. doi: 10.1016/j.eclinm.2023.102036. eCollection 2023 Jun. PMID 37396808